CLINICAL TRIAL: NCT01906645
Title: Care Transitions Innovation (C-TraIn): Study of a Multi-component Transitional Care Intervention for Uninsured and Low-income Publicly Insured Adults
Brief Title: Care Transitions Innovation (C-TraIn)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Honora Englander, Assistant Professor of Medicine, Medical Director of Care Transitions Innovation (C-TraIn), Oregon Health and Science University
Allocation: Randomized | Masking: Single | Purpose: Health Services Research
Other Study IDs: OHSU eIRB 6208
Record Dates: First submitted 2013-07-17; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Hospitalization
Keywords: Patient Readmission; Continuity of Patient Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Usual care consists of 1) a routine nurse intake 2) medication reconciliation performed by treating physicians. Given resource constraints (routine medication reconciliation did not include corroborating medication histories with outpatient pharmacies, routine use of pill cards or pill boxes, or review of Medicaid formularies) Uninsured patients were financially responsible for most medications at discharge. 3) Discharge patient education was performed by inpatient nurses and treating physicians at the time of discharge. 4) Patients without a usual source of primary care were often given a list of the fourteen area safety-net clinics, which have limited capacity for uncompensated care.
- C-TraIn (Experimental): Care Transitions Innovation (C-TraIn) was delivered in addition to usual care, and includes (1) transitional nurse coaching and education, including post-discharge phone calls and home visits for highest risk patients; (2) pharmacy care that includes patient education, medication reconciliation, guidance to inpatient providers to encourage low-cost medications, and provision of 30 days of medications after discharge for those without prescription drug coverage; (3) post-hospital primary care linkages; (4) and explicit efforts at system integration through monthly quality improvement meetings.
  Interventions: Other: Care Transitions Innovation (C-TraIn)

INTERVENTIONS:
Other: Care Transitions Innovation (C-TraIn) — Multi-component transitional care intervention including transitional nursing care, pharmacy care, and medical home linkages
  Arms: C-TraIn

SUMMARY:
The purpose of this protocol is to evaluate the Care Transitons Innovation, a quality improvement project being implemented at OHSU to improve the transition from hospital to home for uninsured and Medicaid patients admitted to general medicine and cardiology wards at OHSU. The evaluation includes a baseline in-person survey and a 30 day post-discharge phone follow-up survey. Prior to C-TraIn, the local healthcare delivery model lacked an effective way to assure timely, safe, and effective follow-up care for uninsured and underinsured hospitalized patients. Most uninsured patients have no source for primary care, and many have limited social support, complex medical problems, and are prescribed many medications. Patients are frequently discharged without any coordinated plan for follow up. Based on a needs assessment performed in 2009 (OHSU eIRB 5514) investigators developed a quality improvement program that will include three major components: 1) a care transitions RN advocate who will see patients in the hospital and after discharge, 2) a pharmacy consultation and 30 days of medications post-discharge, 3) linkages with primary care medical homes, including payment for primary care for uninsured patients who lack a usual source of care, and 4) monthly meetings that serve as a platform for continuous quality improvement. In order to measure the success of our program, investigators will track patient utilization, sociodemographic factors, and patient factors including satisfaction, activation, and self-reported health status. To be included patients must be uninsured, have Oregon Medicaid, or be low income (200% or less of federal poverty level) Medicare recipients, and live within Multnomah, Washington and Clackamas Counties in Oregon.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized on one of seven inpatient treatment teams
* uninsured or low-income publicly insured (Medicaid; Medicare/Medicaid; or Medicare without supplemental insurance and ≤200% poverty level)
* reside in one of three metro-area counties (Multnomah, Washington, Clackamas)

Exclusion Criteria:

* not community dwelling (ie not from a long-term care facility or with plans to discharge to skilled nursing facility)
* no access to a working telephone (participants could list a friend or shelter phone)
* non-English speakding
* HIV positive (HIV+ patients were eligible for overlapping transitional care resources)
* disabling mental illness (as characterized by active psychosis or active suicidal ideation) or severe cognitive deficits
* plans to enter hospice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
30-day hospital readmissions | 30-days
Emergency Department use | 30-days post-discharge

SECONDARY OUTCOMES:
Care Transitions Measure (CTM-3) | Patient report at 30-days post hospital discharge
  The 3 item care transitions measure (CTM-3) is a validated measure that assesses the quality of the care transition. It asks patients to rate agreement with the following:
  1. The hospital staff took my preferences and those of my family or caregiver into account in deciding what my health care needs would be when I left the hospital.
  2. When I left the hospital, I had a good understanding of the things I was responsible for in managing my health.
  3. When I left the hospital, I clearly understood the purpose for taking each of my medications.
  It is being considered by NQF for public reporting. More Background can be found at: http://www.caretransitions.org/documents/CTM_FAQs.pdf
all cause mortality | 30-days post-discharge

OTHER OUTCOMES:
Patient Activation Measure | 30-days post-discharge
  Patient Activation Measure (PAM) is a 13-item validated measure of patient activation developed by Judith Hibbard and colleagues.
  Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the patient activation measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004;39 (4 pt 1):1005-1026.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Englander H, Kansagara D. Planning and designing the care transitions innovation (C-Train) for uninsured and Medicaid patients. J Hosp Med. 2012 Sep;7(7):524-9. doi: 10.1002/jhm.1926. Epub 2012 Mar 12. PMID 22411913
- [Derived] Englander H, Michaels L, Chan B, Kansagara D. The care transitions innovation (C-TraIn) for socioeconomically disadvantaged adults: results of a cluster randomized controlled trial. J Gen Intern Med. 2014 Nov;29(11):1460-7. doi: 10.1007/s11606-014-2903-0. Epub 2014 Jun 10. PMID 24913003